CLINICAL TRIAL: NCT05491902
Title: Pilot PET Study of Regional Cerebral Protein Synthesis in Alzheimer's
Status: Terminated | Type: Observational
Why Stopped: 11C-leucine no longer available at Wolfson Molecular Imaging Centre (after suspension of recruitment due to COVID pandemic)
Sponsor: University of Manchester (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Karl Herholz, Professor and Head of Neuroscience Research at the Wolfson Molecular Imaging Centre, University of Manchester
Other Study IDs: 16/NW/0705
Record Dates: First submitted 2021-09-28; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease
Keywords: [11C]-Leucine; Positron Emission Tomography; Cerebral Protein Synthesis
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early onset mild to moderate AD: Patients aged 50 to 69
  Interventions: Diagnostic Test: [C11] Leucine PET scan; Diagnostic Test: [18F] Flutemetamol PET scan; Diagnostic Test: MRI scan
- Late onset mild to moderate AD: Patients aged 70 and above
  Interventions: Diagnostic Test: [18F] Flutemetamol PET scan; Diagnostic Test: MRI scan
- Older Healthy Volunteer: Aged 50 to 69
  Interventions: Diagnostic Test: [C11] Leucine PET scan; Diagnostic Test: [18F] Flutemetamol PET scan; Diagnostic Test: MRI scan
- Younger Healthy Volunteer: Aged 18 - 25
  Interventions: Diagnostic Test: [C11] Leucine PET scan; Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: [C11] Leucine PET scan — Each participant will receive an i.v. bolus of the PET radioligand, [11C]-Leucine (<100 μg), for each scan. [11C]-Leucine is a PET radioligand has been used and studied clinically (17-23) at micro-doses (<100 μg) with no adverse effects.
  Groups: Early onset mild to moderate AD; Older Healthy Volunteer; Younger Healthy Volunteer
Diagnostic Test: [18F] Flutemetamol PET scan — Each participant will receive an i.v. bolus of the PET radioligand, [18F]-Flutemetamol (< 10 μg), for each scan.
  Groups: Early onset mild to moderate AD; Late onset mild to moderate AD; Older Healthy Volunteer
Diagnostic Test: MRI scan — Scans will be performed on a 1.5T Philips scanner including a 3D T1-weighted scan for co-registration with PET scans and rating of hippocampal atrophy, as well as standard T1 and T2-weighted sequences for rating of white matter lesions.

SUMMARY:
Measuring the rate of cerebral protein synthesis (rCPS) may enable us to better-understand the progression of Alzheimer's Disease (AD). This study is using a new method of measuring rCPS non-invasively, and to offer new approaches to the assessment of new therapeutic strategies in clinical trials.

Previous studies have established the utility of [11C]-Leucine PET to assess the rCPS. This study will use [11C]- Leucine PET to measure rCPS in AD patients versus age-matched and young healthy subjects to determine whether a measurable difference exists.

The study will involve participants receiving up to two PET scans, a structural MRI scan. The PET scanning procedures will involve some withdrawal of blood samples.

The ultimate goal of this proposal is to indicate new routes for treatment of AD.

ELIGIBILITY:
Inclusion Criteria

Patients may be included in the early onset probable AD group if they:

* Are males or females between 50 and 69 years of age, inclusive, with onset of symptoms before age 65;
* Meet the clinical criteria of the National Institute on Aging and the Alzheimer's Association workgroup for probable AD [25]. They have a significant cognitive impairment, Mini Mental State Examination (MMSE) score between 10 and 24 inclusive. Imaging biomarkers (hippocampal volume and cortical amyloid deposition) will be recorded for exploratory correlational analysis with PSR, but will not be used as criteria for inclusion;
* Have a caregiver who can report on their mental status and activities of daily
* living (ADL);
* Must have capacity and be able to give informed consent.
* Willing to comply with protocol and lifestyle restrictions;
* Are women of childbearing potential in whom pregnancy or breast feeding has been excluded by a standard questionnaire (Appendix 3).
* Understanding of English (for questionnaires);
* Participant is ambulant and capable of attending a PET scan visit as an outpatient;
* Participants with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol Section 7.5.1. This criterion must be followed from after the first PET scan until after the follow-up contact;
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test;
* Body weight ≥ 50 kg.

Patients may be included in the late onset probable AD group if they:

* Are males or females ≥70 years of age with onset of symptoms not before age 65;
* Meet the clinical criteria of the National Institute on Aging and the Alzheimer's Association workgroup for probable AD [25]. They have a significant memory impairment, Mini Mental State Examination (MMSE) score between 10 and 24 inclusive. Imaging biomarkers (hippocampal volume and cortical amyloid deposition) will be recorded for exploratory correlational analysis with PSR, but will not be used as criteria for inclusion;
* Have a caregiver who can report on their mental status and activities of daily living (ADL);
* Must have capacity and be able to give informed consent.
* Willing to comply with protocol and lifestyle restrictions;
* Are women of childbearing potential in whom pregnancy or breast feeding has been excluded by a standard questionnaire (appendix).Understanding of English (for questionnaires);
* Participant is ambulant and capable of attending a PET scan visit as an outpatient;
* Participants with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 7.5.1. This criterion must be followed from after the first PET scan until after the follow-up contact;
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test;
* Body weight ≥ 50 kg.

Subjects may be included in the older control group if they:

* Are males or females between 50 and 69 years of age, inclusive;
* Do not have a history of or a current clinically significant neurologic or psychiatric disease and do not have symptoms of cognitive impairment
* Have a Mini Mental State Examination (MMSE) score at screening between 27 and 30, and perform normally on a memory test including delay recall memory;
* Willing to comply with protocol and lifestyle restrictions;
* Are women of childbearing potential in whom pregnancy or breast feeding has been excluded by a standard questionnaire (appendix).Understanding of English (for questionnaires);
* Participant is ambulant and capable of attending a PET scan visit as an outpatient;
* Participants with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 7.5.1. This criterion must be followed from after the first PET scan until after the follow-up contact;
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test;
* Body weight ≥ 50 kg.

Subjects may be included in the young control group if they:

* Are males or females between 18 and 25 years of age, inclusive;
* Do not have a history of or a current clinically significant neurologic or psychiatric disease and do not have symptoms of cognitive impairment;
* Do not have a first grade relative with early onset AD;
* Have a Mini Mental State Examination (MMSE) score at screening between
* 27 and 30, and perform normally on a memory test including delay recall memory;
* Willing to comply with protocol and lifestyle restrictions;
* Are women of childbearing potential in whom pregnancy or breast feeding has been excluded by a standard questionnaire (appendix).Understanding of English (for questionnaires);
* Participant is ambulant and capable of attending a PET scan visit as an outpatient;
* Participants with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 7.5.1. This criterion must be followed from after the first PET scan until after the follow-up contact;
* Adequate collateral flow to the radial and ulnar arteries in both hands as determined by an Allen's test;
* Body weight ≥ 50 kg.

Exclusion Criteria:

* Have a history of or a current clinically significant neurologic or psychiatric disease (other than AD);
* Have a current clinically significant endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer;
* Have a clinically significant infectious disease, including Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV) infection;
* Have a recent history of alcohol or substance abuse or dependence;
* Clinically significant brain injury or abnormality, other than associated with AD;
* Are women of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using reliable methods of contraception (as detailed in Section 7.5.1);
* Treatment with stable doses of psychotropic medication is not prohibited. In particular, patients with AD may be on a stable dose of an anticholinesterase, memantine, neuroleptic or antidepressant, and may be taking vitamin E at the time of imaging;
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
* History of or suffers from claustrophobia or participant feels unable to lie flat and still on their back for a period of up to 90 minutes in the PET scanner;
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations or occupational exposure in the past 12 months or greater than 10 mSv in a single year including the proposed study. Clinical exposure from which the participant receives a direct benefit is not included in these calculations;
* Previous inclusion in a research and/or medical protocol involving study medication within the last 3 months;
* In the opinion of the study team they are unlikely to comply with the study protocol and restrictions that it imposes. ;
* Contraindications for participants undergoing an MRI scan (including but not limited to metal implants pacemakers, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 12 AD participants will be recruited by the Salford Royal Foundation Trust in collaboration with clinical partners in appropriate clinical services for dementia. Up to 12 healthy controls will be recruited by approaching spouses and carers of patients or through the "Join Dementia Research" and "Citizen Scientist Salford" networks.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Regional changes in Protein Synthesis Rate in AD brain compared to age-matched controls | 2 years after completion of patient recruitment
  A primary outcome of this study will be to determine if regional changes in PSR, as measured by [11C]-Leucine PET, in early onset AD brain are lower compared to age-matched controls. The output parameter used to determine this will be derived from the most appropriate PET pharmacokinetic model for this ligand in human.
Regional changes in Protein Synthesis Rate in healthy controls | 2 years after completion of patient recruitment
  Comparison of any regional changes in PSR from the CNS of young healthy controls with older healthy controls, will occur, to assess if there is an age-dependent decline in PSR in healthy human brain and whether its regional distribution is different from disease-related changes.

SECONDARY OUTCOMES:
Regional changes in Protein Synthesis Rate in AD patients | 2 years after completion of patient recruitment
  Comparison of any regional changes in PSR from the CNS of early onset AD patients compared with late onset AD patients.Assessment of amyloid deposition effect on rCPS.

OTHER OUTCOMES:
Meta-analysis | 2 years after completion of patient recruitment
  Meta-analysis of data collected from this study with existing literature data-sets to (1) increase the overall number of comparable data-sets which would allow for further statistical evaluation of these datasets with these higher n-numbers, and (2) to assess the consistency of data collected between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Wolfson Molecular Imaging Centre (University of Manchester), Manchester
  - Salford Royal NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No